CLINICAL TRIAL: NCT02170636
Title: Bioavailability of BIBR 953 ZW After 50 mg of BIBR 1048 MS (Oral Prodrug of BIBR 953) in 4 Experimental Formulations Relative to Drinking Solution of BIBR 1048 MS, Each Treatment Given Bid Over 3 Days, in Healthy Subjects. Intraindividual Comparison (5-way Crossover), Randomised, Open. For Each of the 5 Treatments, Investigation of 2 Conditions: With and Without Pantoprazole (Intraindividual, Open Comparison).
Brief Title: Bioavailability of BIBR 953 ZW After Oral Administration of BIBR 1048 MS in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.32
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (2):
- Period 1: BIBR 1048 MS + Pantoprazole (Experimental): Five treatments with oral administration of 50 mg BIBR 1048 MS (bid for 3 days) and 40 mg Pantoprazole (bid). Randomised sequence.
  BIBR 1048 MS Capsule E with pantoprazole; BIBR 1048 MS Capsule F with pantoprazole; BIBR 1048 MS Capsule G with pantoprazole; BIBR 1048 MS Tablet H with pantoprazole; BIBR 1048 MS Drinking solution with pantoprazole
  Interventions: Drug: BIBR 1048 MS Capsule E; Drug: BIBR 1048 MS Capsule F; Drug: BIBR 1048 MS Capsule G; Drug: BIBR 1048 MS Tablet H; Drug: BIBR 1048 MS Drinking solution; Drug: Pantoprazole
- Period 2: BIBR 1048 MS (Experimental): Three treatments (fixed sequence) with oral administration of 50 mg BIBR 1048 MS (bid for 3 days).
  1. BIBR 1048 MS Capsule E without pantoprazole;
  2. BIBR 1048 MS Tablet H without pantoprazole;
  3. BIBR 1048 MS Drinking solution without pantoprazole
  Interventions: Drug: BIBR 1048 MS Capsule E; Drug: BIBR 1048 MS Tablet H; Drug: BIBR 1048 MS Drinking solution

INTERVENTIONS:
Drug: BIBR 1048 MS Capsule E — 50 mg BIBR 1048 MS
Drug: BIBR 1048 MS Capsule F — 50 mg BIBR 1048 MS
  Arms: Period 1: BIBR 1048 MS + Pantoprazole
Drug: BIBR 1048 MS Capsule G — 50 mg BIBR 1048 MS
  Arms: Period 1: BIBR 1048 MS + Pantoprazole
Drug: BIBR 1048 MS Tablet H — 50 mg BIBR 1048 MS
Drug: BIBR 1048 MS Drinking solution — 50 mg BIBR 1048 MS tartaric acid solution
Drug: Pantoprazole — 40 mg Pantoprazole
  Arms: Period 1: BIBR 1048 MS + Pantoprazole

SUMMARY:
Study to assess the amount of BIBR 953 ZW in urine after administration of 50 mg BIBR 1048 bid over three days each administered as four experimental formulations relative to drinking solution with and without coadministration of 40 mg Pantoprazole

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 55 years
* Broca ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2002-01; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Total amount of BIBR 953 ZW excreted into urine over one dose interval (Ae0-12) | Day 1 to 16 of each treatment period
AUCss (area under the plasma concentration-time curve at steady state) of BIBR 953 ZW | 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after administration of study drug on day 3 of second treatment period

SECONDARY OUTCOMES:
Cmax,ss (maximum concentration at steady state) of BIBR 953 ZW | 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after administration of study drug on day 3 of second treatment period
tmax,ss (time from dosing to Cmax at steady state) of BIBR 953 ZW | 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours after administration of study drug on day 3 of second treatment period